CLINICAL TRIAL: NCT05673070
Title: Use of Ritual Prenatal Multivitamins to Improve Nutrition Status and Health Outcomes During Pregnancy
Brief Title: Use of Ritual Prenatal Multivitamins for Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Xinyin Jiang, Associate professor, City University of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-0670-Brooklyn
Record Dates: First submitted 2022-12-06; First posted 2023-01-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related; Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: Prenatal arm: pregnant women at gestational week 12-14 will be randomized to either receive a Ritual prenatal MVI (n=35) or a control commercially available prenatal MVI (n=35) through out pregnancy
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the investigators will know the group assignment. Supplements will be prepared by the pharmacy and marked with randomly generated ID numbers. Grouping will be revealed by pharmacy at end of the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ritual Epre (Experimental): This group will receive 2 Ritual Epre multivitamin-mineral supplement pills daily.
  Interventions: Dietary Supplement: Ritual Epre Multivitamin-mineral supplement
- Control MVI (Active Comparator): For the prenatal arm, this group will receive a control multivitamin-mineral supplement pill and a 200 mg docosahexaenoic acid (DHA) pill that are commercially available.
  Interventions: Dietary Supplement: control MVI

INTERVENTIONS:
Dietary Supplement: Ritual Epre Multivitamin-mineral supplement — The Ritual Epre supplement uses methyl folate instead of folic acid and has higher vitamin D and biotin contents compared to the control supplement.
  Arms: Ritual Epre
Dietary Supplement: control MVI — The control MVI supplement is a commercially available product from another brand. Since this MVI doesn't contain DHA, a pill of DHA will also be provided to participants in this group.
  Arms: Control MVI

SUMMARY:
Prenatal multivitamin/multimineral supplements (MVI) provide important nutrition supplement to the diet of pregnant women to cover potential deficiencies and optimize nutrition status of both mom and baby, especially when the diet is suboptimal or nutrient demand is high while absorption is hindered by various factors such as genetic variance and gastrointestinal function. In this double-blind, randomized, controlled trial, the investigators will recruit 70 pregnant women at gestational week 12-14 and randomly assign them to either receive a Ritual prenatal MVI (n=35) or another commercially available prenatal MVI (n=35) through out pregnancy. Both supplements are over the counter and commercially available. The major differences between the two MVIs are the chemical form of folate as either 5-methyl-tetrahydrofolate or folic acid, and the dosages of vitamin D, biotin, and docosahexaenoic acid. The investigators will collect blood samples in each trimester of pregnancy and the placenta and cord blood at delivery to assess differences in blood nutrient levels. The investigators hypothesize that consumption of Ritual MVI leads to better nutrition status and biomarkers in maternal-fetal dyads compared to control during the antepartum period.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women are qualified to participate if they are over 18 years of age, having singleton pregnancy, and without any of the conditions listed in the exclusion criteria.

Exclusion Criteria:

* Exclusion criteria include diabetes, cardiovascular conditions and liver disease prior to and during pregnancy because these diseases affect metabolism of several nutrients and thus may lead to differences in the MVI intake and nutrient status relationship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Folate status | after 24 weeks of intervention
  The investigators hypothesize that the group that consumes Ritual would have less unmetabolized folic acid in the blood than the control group. A greater proportion of participants would have supranutritional levels of folate (> 20 ng/mL serum folate) in the control versus Ritual group.
Biotin status | after 24 weeks of intervention
  The investigators hypothesize that the group that consumes Ritual would have higher levels of biotin and lower levels of 3-HIA and 3-HIA-carnitine in the maternal and cord blood than the control group.
vitamin D status | after 24 weeks of intervention
  The investigators hypothesize that the group that consumes Ritual would have higher levels of vitamin D metabolites in the maternal and cord blood than the control group.
placental functional gene expression regulation | after 24 weeks of intervention
  The investigators hypothesize that the group that consumes Ritual would have higher expression of vitamin D response genes and lower expression of inflammatory and stress genes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brooklyn College of City University of New York, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No